CLINICAL TRIAL: NCT05021003
Title: Effects of Core Stabilization Training With and Without Pressure Biofeedback in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0117 Hashim
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain
Keywords: Pain; Back; Core stabilization; Pressure biofeedback
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): : Core stabilization training with pressure biofeedback unit
  Interventions: Other: pressure biofeedback
- Group B (Active Comparator): : Core stabilization training without pressure biofeedback unit
  Interventions: Other: core stabilization exercises

INTERVENTIONS:
Other: pressure biofeedback — : Core stabilization training with pressure biofeedback unit
  Arms: Group A
Other: core stabilization exercises — : Core stabilization training without pressure biofeedback unit
  Arms: Group B

SUMMARY:
Mechanical low back pain is an impairment of musculoskeletal system. Lifetime prevalence of low back pain is 60-85%. Frequent micro-trauma to the structures of the spine, poor control and stabilization leads to LBP and eventually causes functional limitation. The objective of the study to find whether Core Stabilization Training with Pressure Biofeedback could reduce pain and improves functional activity in patients with mechanical low back pain. To study the effectiveness of Core Stabilization Training with Pressure Biofeedback in reducing pain and improving functional activity in subjects with mechanical low backpain between the age group of 25-40 years. To find out the effect of core stabilization training with pressure biofeedback in reducing pain and improving functional activity in subjects with mechanical low back pain between the age group of 25-40 years. The study will be conducted on 30 subjects between the age group of 25-40 years with mechanical low back pain and according to the inclusion criteria were recruited in the study. NPRS at rest and activity, Modified ODI will assess PRE and POST treatment. P value: less than 0.05 using SPSS (Statistical package for social sciences) for NPRS(pain at rest and activity) and modified ODI i.e. core stabilization training with pressure biofeedback had statistical improvement in NPRS (Pain at rest and activity) and modified ODI score. Core stabilization training with pressure biofeedback is effective inreducing pain (at rest and activity) and functional disability in subjects between the age group of 25-40 years with mechanical low back pain

ELIGIBILITY:
Inclusion Criteria:\

* Male and female patients between the age group 25-40 years having mechanical low back pain persisting for at least 6 months upto1 year.
* Patients complaining Pain when sitting or standing for a long period or Pain when driving long distance, getting in and out of the car or lifting activities.
* Patients with minimum and moderate disability based on Modified Oswestry Disability Index (ODI).
* Patients with greater than and equal to 7 score on NPRS.

Exclusion Criteria:

* Structural deformity (scoliosis, lordosis).
* Systematic inflammatory disease (vasculitis, connective tissue disease and granulomatous disease).
* Nerve root compression (Disc bulge and Lumbar radiculopathy).
* History of spinal surgery or fractures (laminectomy).

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 4 weeks
  In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity [1]. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible
oswestry disability index | 4 weeks
  Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burton AK, Balague F, Cardon G, Eriksen HR, Henrotin Y, Lahad A, Leclerc A, Muller G, van der Beek AJ; COST B13 Working Group on Guidelines for Prevention in Low Back Pain. Chapter 2. European guidelines for prevention in low back pain : November 2004. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S136-68. doi: 10.1007/s00586-006-1070-3. No abstract available. PMID 16550446
- [Background] Carlsson AM. Assessment of chronic pain. I. Aspects of the reliability and validity of the visual analogue scale. Pain. 1983 May;16(1):87-101. doi: 10.1016/0304-3959(83)90088-X. PMID 6602967
- [Background] Bhadauria EA, Gurudut P. Comparative effectiveness of lumbar stabilization, dynamic strengthening, and Pilates on chronic low back pain: randomized clinical trial. J Exerc Rehabil. 2017 Aug 29;13(4):477-485. doi: 10.12965/jer.1734972.486. eCollection 2017 Aug. PMID 29114516